CLINICAL TRIAL: NCT04133584
Title: Multiple Centers, Randomized, and Control Trail on the Immunogenicity and Safety of the Simultaneously Vaccination of Inactivated Enterovirus 71 Vaccine (EV71) and Seasonal Influenza Vaccine(SIV)
Brief Title: The Immunogenicity and Safety of the Vaccination of Inactivated Enterovirus 71 Vaccine and Seasonal Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Collaborators: China National Biotec Group Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZJCDC20190918
Record Dates: First submitted 2019-09-18; First posted 2019-10-21 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Seasonal Influenza; Hand, Foot and Mouth Disease
Keywords: Immunogenicity; Safety; Enterovirus 71 Vaccine; seasonal influenza vaccine
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 EV71 +SIV (Experimental): Give 2 doses of Inactivated Enterovirus 71 Vaccine (EV71) and seasonal influenza vaccine(SIV) simultaneously with 28 days apart
  Interventions: Biological: EV71 +SIV
- Group 2 EV71 (Active Comparator): Give 2 doses of Inactivated Enterovirus 71 Vaccine (EV71) with 28 days apart
  Interventions: Biological: EV71
- Group 3 SIV (Active Comparator): Give 2 doses of seasonal influenza vaccine(SIV) simultaneously with 28 days apart
  Interventions: Biological: SIV

INTERVENTIONS:
Biological: EV71 +SIV — Give 2 doses of EV71 +SIV, get 2 blood samples before the first dose and 28-43 days after the last dose.
  Arms: Group 1 EV71 +SIV
Biological: EV71 — Give 2 doses of EV71 , get 2 blood samples before the first dose and 28-43 days after the last
  Arms: Group 2 EV71
Biological: SIV — Give 2 doses of SIV , get 2 blood samples before the first dose and 28-43 days after the last
  Arms: Group 3 SIV

SUMMARY:
The purpose of this study is to evaluate the Immunogenicity and safety of the simultaneously vaccination of Inactivated Enterovirus 71 Vaccine (EV71) and seasonal influenza vaccine(SIV)

DETAILED DESCRIPTION:
Main subjects:

The seroconversion rate for each antigen when EV71 is administrated with SIV

Secondary subjects:

The positive rate of antibody for each antigen when EV71 is administrated with SIV The safety for each antigen when EV71 is administrated with SIV

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal acceptable representative is willing and able to understand the protocol requirements and provide informed consent.
* Participant is aged ≥ 6 month to <12 months.
* Participant without preventive inoculation of Enterovirus 71 Vaccine ,seasonal influenza vaccine vaccine and previous history of Enterovirus.
* Subject and parent/guardian able to attend all scheduled visits and comply with all trial procedures.
* Body temperature ≤ 37.0#.

Exclusion Criteria:

* Known allergy to any constituent of the vaccine.

  * Known acute illness, severe chronic disease, acute exacerbation of chronic disease and fever.
  * Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth.
  * Reported the history of allergies, convulsions, epilepsy, mental illness and brain disease and clear serious systemic reaction.
  * Known bleeding disorder.
  * Receipt of the whole blood, blood plasma or immunoglobulin before the trial vaccination.
  * Reported the history of acute illness had need systemic antibiotics or antiviral treatment of infections in the 7 days preceding the trial vaccination.
  * An acute illness with or without fever (temperature ≥ 38.0#) in the 3 days preceding enrollment in the trial.
  * Participation in any other intervention clinical trial.
  * Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the vaccine.

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1134 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
immunogenicity evaluation | change from baseline antibody concentration at 28 days after the last dose
  The positive rate of antibody

SECONDARY OUTCOMES:
safety evaluation: The occurrence of adverse events | up to 30 days after every injection
  The occurrence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Liandu Center for Disease Control and Prevention, Lishui, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No